CLINICAL TRIAL: NCT06873841
Title: Can the Cognitive-Psychophysiological Treatment of Tics be Optimized Through Biofeedback in Adolescents and Emerging Adults With Tourette Syndrome? - A Randomized Clinical Trial
Brief Title: Cognitive-psychophysiological Treatment for Tics in Young People With Tourette's Syndrome With or Without Biofeedback
Acronym: CoBRa
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université du Québec a Montréal (Other)
Collaborators: Ciusss de L'Est de l'Île de Montréal (Other)
Responsible Party: Principal Investigator, Julie Leclerc, Full professor, psychology department, UQAM. Researcher & Mental Health Research Director, Centre intégré universitaire santé et services sociaux (CIUSSS) Nord-de-l'Île-de-Montréal. Associate Researcher, Institut Universitaire Santé Mentale de Montreal, Université du Québec a Montréal
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PJT-191682
Record Dates: First submitted 2025-01-21; First posted 2025-03-13 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Tourette Syndrome; Tics; Tourette Syndrome in Adolescence
Keywords: CoPs; Biofeedback; cognitive-psychophysiological therapy; Tourette; Young adults; Tics; Treatment
MeSH Terms: conditions — Tourette Syndrome; Tics | interventions — Biofeedback, Psychology

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Randomization ensures that participants will not immediately know their treatment modality. However, since we do not have a drug under study and the interventions are therapies, the participant may end up knowing their group by themselves. To avoid biases, the evaluators will have no idea which group the participant belongs to. Only the therapists will know the participants' modality, as they are the ones who will administer it.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive-psychophysiological therapy (CoPs). (Active Comparator): Six therapeutic steps: 1) Awareness training; 2) Profile of high/low-risk situations for tics; 3) Muscular discrimination; 4) Reduction of sensorimotor activation and modification of action planning style; 5) Cognitive, metacognitive, and behavioral restructuring in high-risk tic situations; 6) Generalization and relapse prevention.
  The individual sessions last 80 minutes: 55 minutes of therapy, 20 minutes of active listening and 5 minutes for a computer activity. The active listening and activity are unrelated to the analyses but ensure that treatment modalities are equivalent in duration and use of a computer. Participants will be informed about the duration of the therapy (10 to 12 sessions weekly) and that its completion requires continuous attendance at the sessions. The program has been adapted for youth with a treatment guide containing examples and exercises tailored for better understanding. Adolescents aged 14 to 17 will receive this manual to support their comprehension.
  Interventions: Behavioral: Cognitive psychophysiological
- Cognitive-psychophysiological therapy (CoPs) combined with biofeedback exercises. (Experimental): After each 55-minute CoPs session (same protocol as arm 1), 25 minutes will be dedicated to biofeedback exercises (80 minutes total). This 25-minute period includes 2 minutes to record the baseline resting level, 15 minutes for the active biofeedback session, and 2 minutes for the second resting measurement.
  Active electromyographic (EMG) biofeedback will take the form of computer-generated graphs displayed on a screen at 2 meters (horizontal angle). Changes in muscle activity will cause the movement of a balance with a silvered ball; the graphical feedback of this stimulus is particularly effective in capturing the participant's attention and interactive engagement. The goal is to contract the arm muscle to keep the ball balanced for 5 minutes for each arm, then 5 minutes with both arms (15 minutes).
  Interventions: Behavioral: Cognitive psychophysiological and Biofeedback

INTERVENTIONS:
Behavioral: Cognitive psychophysiological — Focus on the processes influencing thoughts and behaviors underlying tics.
  Arms: Cognitive-psychophysiological therapy (CoPs).
Behavioral: Cognitive psychophysiological and Biofeedback — Biofeedback refers to visual exercises that help improve movement control.
  Arms: Cognitive-psychophysiological therapy (CoPs) combined with biofeedback exercises.

SUMMARY:
The goal of this clinical trial is to compare the effectiveness of CoPs therapy with or without the therapeutic component of biofeedback in treating tics in Tourette Syndrome with emerging young adults.

Hypotheses:

1. The CoPs+Biofeedback treatment will improve the severity of tics (YGTSS) and the Clinical Global Impression, surpassing the clinical significance threshold of CoPs treatment alone.
2. We expect that the identified variables (psychosocial, neurocognitive, biological) will predict the improvement of tics.

Researchers will compare if the biofeedback treatment will improve the severity of tics.

* In the pre-test, participants will undergo two interviews, each lasting 3 hours. These interviews will assess (through a battery of tests) the severity of tics as well as the psychosocial, biological, and neurocognitive aspects of functioning. A general assessment of intelligence and executive functions will also be conducted.
* They will next attend 10 to 12 therapy sessions, with or without biofeedback. (The biofeedback component is explained in more detail in the ''Study Design'' section).
* The post-test follow-ups consist of two evaluations: one 3 months after the end of the treatment and the other 6 months after. The evaluation will be done using the same battery of tests as during the pre-test interview.

DETAILED DESCRIPTION:
* The project explanations are in English for everyone's ease of understanding, but our study is conducted in French. *

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of TS or to experience bothersome tics;
* Be aged 14 to 21 years inclusive at the start of therapy.

Exclusion Criteria:

* Present a sensorimotor impairment;
* Have a diagnosis of intellectual disability (intelligence quotient below 75);
* Alcohol or drug abuse;
* A neurological issue (e.g., hemifacial spasms, Huntington's disease);
* Change medication one month or less before step 1 and up to step 4 (last measurement time) without informing a member of the research team;
* Simultaneously receive another intervention for tics (e.g., psychologist, massage therapist) without informing a research team member.

Ages: 14 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Primary outcome | The YGTSS is administered trough the study completion, an average of 1 year (T1 pre, T2 post, T3 follow up (3 months), T4 follow up (6 months))
  The Yale Global Tic Severity Scale (YGTSS) provides an assessment of motor and vocal tics based on 5 dimensions: number, frequency, intensity, complexity, and interference. A subtotal of 50 is used to determine the severity of the tics. A separate scale assesses impairment, or the overall effect of tic disorders on daily functioning, with another subtotal of 50. In this study, only the tic severity score out of 50 will be used (comparable to other studies focusing on tics).

SECONDARY OUTCOMES:
Conners | Administered trough study completion, an average of 1 year (T1 pre, T2 post, T3 follow up (3 months), T4 follow up (6 months)).
  Psychosocial measures For ADHD symptoms, the Conners 3 (8-18 years) or Conners' Adult ADHD Rating Scales (CAARS)
CY-BOCS | Administered trough study completion, an average of 1 year (T1 pre, T2 post, T3 follow up (3 months), T4 follow up (6 months)).
  For OCD symptoms, the Yale-Brown Obsessive-Compulsive Scale (CY-BOCS)
STAI | Administered trough study completion, an average of 1 year (T1 pre, T2 post, T3 follow up (3 months), T4 follow up (6 months)).
  For anxiety symptoms, the State-Trait Anxiety Inventory (STAI).
Perfectionism Scale | Administered trough study completion, an average of 1 year (T1 pre, T2 post, T3 follow up (3 months), T4 follow up (6 months)).
  The adapted/inadapted Perfectionism Scale
Beck Depression Invetory | Administered trough study completion, an average of 1 year (T1 pre, T2 post, T3 follow up (3 months), T4 follow up (6 months)).
  For mood-related symptoms, the Beck Depression Inventory will be used.
STOP | Administered trough study completion, an average of 1 year (T1 pre, T2 post, T3 follow up (3 months), T4 follow up (6 months)).
  The Style of Planning Action (STOP)
Self-Esteem Inventory | Administered trough study completion, an average of 1 year (T1 pre, T2 post, T3 follow up (3 months), T4 follow up (6 months)).
  The short version of the Self-Esteem Inventory.
TS-Quality of Life Scale | Administered trough study completion, an average of 1 year (T1 pre, T2 post, T3 follow up (3 months), T4 follow up (6 months)).
  TS-Quality of Life Scale will also be used.
Perdue Pegboard Test | Administered trough study completion, an average of 1 year (T1 pre, T2 post, T3 follow up (3 months), T4 follow up (6 months)).
  The evaluation of fine motor dexterity using the Purdue Pegboard will determine the baseline equivalence between groups and test functional differences after treatment. The Finger-Tapping Test will be administered to assess speed and motor control.
Perceived Stress Scale (PSS-14) | Administered trough study completion, an average of 1 year (T1 pre, T2 post, T3 follow up (3 months), T4 follow up (6 months)).
  We will collect a hair sample to measure the cortisol levels of the participants: a 14-item Perceived Stress Scale (PSS-14) will be administered at the 4 time points of measurement.
Finger-Tapping Test | Administered trough study completion, an average of 1 year (T1 pre, T2 post, T3 follow up (3 months), T4 follow up (6 months)).
  The Finger-Tapping Test will be administered to assess speed and motor control.
DKEFS CWIT | Only in T1 (pre-test) , up to 4 weeks ( first interview).
  Participants will be assessed with the 4 sections of the DKEFS CWIT: color naming, word reading, inhibition.
Brief Cannabis Consumption Questionnaire | Only in T1 (pre-test) , up to 4 weeks ( first interview).
  To attest the consumption of cannabis.

OTHER OUTCOMES:
SCID-5-RV130 | Only in T1 (pre-test) , up to 4 weeks ( first interview).
  The Structured Clinical Interview for DSM-5 - Research (SCID-5-RV130) will allow for clinical screening of disorders that may present a differential or comorbid diagnosis with PTSD, which could impact treatment engagement or outcomes.
BASC-3-SRP131 | Only in T1 (pre-test) , up to 4 weeks ( first interview).
  The Behavioral Assessment System, 3rd Edition - Self-Report of Personality (BASC-3-SRP131) will be administered to provide an overall profile of affect and behavior, complementing the SCID-5-RV.
Bem Sex Role | Only in T1 (pre-test) , up to 4 weeks ( first interview).
  Sex assigned at birth and gender identity will be assessed using the Bem Sex Role Inventory.
Wechsler | Only in T1 (pre-test) , up to 4 weeks (first interview).
  General intelligence will be evaluated through subscales of the Wechsler Intelligence Scale for Children/Adults, depending on the participant's age (WAIS-IV, WISC-V: Vocabulary, Matrices).
BRIEF | Only in T1 (pre-test) , up to 4 weeks ( first interview).
  Executive functions will also be screened using the Brief Inventory of Executive Function (BRIEF), (version for ages 14-18 years or adults).

CONTACTS AND LOCATIONS:
Overall Officials: Julie Leclerc, Psychology, Principal Investigator — Université du Québec à Montréal- UQAM; Marc Lavoie, Psychology, Study Chair — Université TÉLUQ; Marie-France Marin, Psychology, Study Chair — Université du Québec à Montréal-UQAM
Locations (1):
- Centre intégré universitaire de santé et de services sociaux du Nord-de-l'Île-de-Montréal, Hôpital Rivières-des-Prairies, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No